CLINICAL TRIAL: NCT01608958
Title: Intravenous and Intramuscular Administration of Oxytocin in the Third Stage of Labor for Prevention of Postpartum Hemorrhage
Brief Title: IV vs IM Oxytocin in the Third Stage of Labor for Prevention of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Center for Research and Consultancy in Reproductive Health (Other); Huong Vuong Hospital (Unknown); MOH Etlik Zubeyde Hanim Women's Health Training and Research Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3000
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; Oxytocin; Third stage of labor; Hemoglobin; Prevention; Intravenous; Intramuscular
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV infusion (Active Comparator): Oxytocin 10 IU will be administered IV infusion according to randomization assignment as soon as possible after delivery of the baby.
  Interventions: Drug: Oxytocin
- IM Injection (Active Comparator): Oxytocin 10 IU will be administered IM according to randomization assignment as soon as possible after delivery of the baby.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — 10 IU oxytocin in 500 ml infusion
  Arms: IV infusion
Drug: Oxytocin — 10 IU oxytocin IM injection
  Arms: IM Injection

SUMMARY:
The study will evaluate whether prophylactic oxytocin administered in the third stage of labor via IV infusion results in a lower mean blood loss compared to IM injection.

DETAILED DESCRIPTION:
The study will compare the effect of IV infusion and IM oxytocin administration on the proportion of women who experience blood loss greater than or equal t 350 ml, the proportion of women who experience blood loss greater than or equal to 500 ml, side effects, adverse events and change in hemoglobin pre- to post-delivery. It will also assess whether a bleeding history questionnaire can identify women at risk for excessive bleeding and help to define the distribution of bleeding scores among women with and without excessive bleeding.

ELIGIBILITY:
Inclusion Criteria:

* All women who present in active labor for a live birth at the study hospital will be considered for participation in the study

Exclusion Criteria: Women who are:

* Planned or transferred for delivery via Cesarean section
* Not delivering a live birth
* Unable to provide informed consent due to mental impairment, distress during labor or other reason
* Unwilling and/or unable to respond to questionnaires about background characteristics and/or bleeding history.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean blood loss (ml) | minimum of 1 hour after delivery of baby

SECONDARY OUTCOMES:
Proportion of women who bleed greater or equal to 350 ml, 500 ml and 1000 ml | minimum of 1 hour after delivery of baby
Change in hemoglobin from pre-delivery to postpartum | 12-24 hours after delivery
  Post-delivery hemoglobin using a Hemocue® Hemoglobin machine + cuvette will be taken at least 24 after delivery and before the woman leaves the facility. If the woman has received IV fluids, hemoglobin will be measured at least 12 hours after removal of the IV prior to discharge.
Time to placental delivery | minimum of 1 hour after delivery of baby
Administration of additional oxytocin, other uterotonics, or other interventions such as blood transfusion and hysterectomy | minimum of 1 hour after delivery of baby
Side effects 1 hour postpartum | 1 hour postpartum
Bleeding scores calculated from a standardized questionnaire administered on arrival to labor ward | arrival to labor ward

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Ilana Dzuba, MHS, Principal Investigator — Gynuity Health Projects; Jill Durocher, Principal Investigator — Gynuity Health Projects; Jennifer Blum, MPH, Principal Investigator — Gynuity Health Projects
Locations (3):
- Hospital Gineco-Obstétrico Isidro Ayora, Quito, Ecuador
- SB Etlik Zübeyde Hanım Kadın Hastalıkları Eğitim ve Araştırma Hastanesi, Ankara, Turkey (Türkiye)
- Huong Vuong Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Oladapo OT, Okusanya BO, Abalos E, Gallos ID, Papadopoulou A. Intravenous versus intramuscular prophylactic oxytocin for the third stage of labour. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD009332. doi: 10.1002/14651858.CD009332.pub4. PMID 33169839